CLINICAL TRIAL: NCT03467945
Title: Randomized, Open Label, Single Dose, 4 Treatment, 4 Period, Crossover Design (4 x 4) Trial to Evaluate the Bioequivalence and Secondarily Drug - Drug Interaction of Fixed Combination of Metformin Tablets 1000 mg/Gliclazide 30 mg MR, Compared With the Co-administration of Individual Tablets and Individual Administration of Each Single Tablet (Metformin 1000 mg XR and Gliclazide 30 mg MR) in Healthy Volunteers
Brief Title: Bioequivalence and Drug - Drug Interaction Study of Metformin/Gliclazide in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EMR200763_003
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Metformin; Gliclazide; Bioequivalence; Drug-drug Interaction; Pharmacokinetics
MeSH Terms: interventions — Metformin; Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Participants received single oral dose of metformin 1000 milligram (mg) and gliclazide 30 mg fixed combination tablet in treatment period 1 followed by concomitant oral dosing of metformin 1000 mg and gliclazide 30 mg in treatment period 2 followed by single oral dose of metformin 1000 mg in treatment period 3 and then a single oral dose of gliclazide 30 mg in treatment period 4. Each treatment period was separated by a 14-day wash-out period.
  Interventions: Drug: Metformin/Gliclazide Fixed Combination; Drug: Metformin; Drug: Gliclazide
- Treatment Sequence 2 (Experimental): Participants received concomitant oral dosing of metformin 1000 mg and gliclazide 30 mg in treatment period 1 followed by single oral dose of gliclazide 30 mg in treatment period 2 followed by single oral dose of metformin 1000 mg and gliclazide 30 mg fixed combination tablet in treatment period 3 and then single oral dose of metformin 1000 mg in treatment period 4. Each treatment period was separated by a 14-day wash-out period.
  Interventions: Drug: Metformin/Gliclazide Fixed Combination; Drug: Metformin; Drug: Gliclazide
- Treatment Sequence 3 (Experimental): Participants received single oral dose of metformin 1000 mg in treatment period 1 followed by single oral dose of metformin 1000 mg and gliclazide 30 mg fixed combination tablet in treatment period 2 followed by single oral dose of gliclazide 30 mg in treatment period 3 and then concomitant oral dosing of metformin 1000 mg and gliclazide 30 mg in treatment period 4. Each treatment period was separated by a 14-day wash-out period.
  Interventions: Drug: Metformin/Gliclazide Fixed Combination; Drug: Metformin; Drug: Gliclazide
- Treatment Sequence 4 (Experimental): Participants received single oral dose of gliclazide 30 mg in treatment period 1 followed by single oral dose of metformin 1000 mg in treatment period 2 followed by concomitant oral dosing of metformin 1000 mg and gliclazide 30 mg in treatment period 3 and then single oral dose of metformin 1000 mg and gliclazide 30 mg fixed combination tablet in treatment period 4. Each treatment period was separated by a 14-day wash-out period.
  Interventions: Drug: Metformin/Gliclazide Fixed Combination; Drug: Metformin; Drug: Gliclazide

INTERVENTIONS:
Drug: Metformin/Gliclazide Fixed Combination — Participants received single oral dose of Metformin and Gliclazide fixed combination tablet in treatment period 1, 2, 3 or 4.
Drug: Metformin — Participants received single oral dose of Metformin tablet in treatment period 1, 2, 3 or 4.
Drug: Gliclazide — Participants received single oral dose of Gliclazide tablet in treatment period 1, 2, 3 or 4.

SUMMARY:
This study investigated the bioequivalence and drug-drug interaction of Metformin/Gliclazide fixed combination tablet compared to co-administration of individual tablets of Metformin and Gliclazide.

ELIGIBILITY:
Inclusion Criteria:

* Participants has given written informed consent before any study-related activities were carried out
* Ethnic origin: Mexicans
* Weight between 55 and 95 kilogram (kg)
* Body mass index between 18.5 and 27 kilogram per meter square (kg/m^2)
* Not smoking more than 5 cigarettes or 1 cigar or 1 pipe per day (or non smokers)
* Good physical and mental health status
* Vital signs (blood pressure and pulse) in supine position within the normal range or showing no clinically relevant deviation as judged by the Investigator
* Electrocardiogram recording (12-lead) without signs of clinically relevant pathology in particular QTc (Bazett) <450 milliseconds (ms)
* All values for biochemistry and hematology tests of blood and urine within the normal range or showing no clinically relevant deviation as judged by the Investigator
* All women of childbearing potential (WOCBP) were not nursing, were not pregnant, and were using highly effective methods of birth control for a period of at least one month before and after dosing
* All women of childbearing potential must have negative tests for pregnancy at screening, and at day -1 for each treatment period and at end of trial (EOT)
* Negative screen for alcohol and drugs of abuse at Screening and on each admission
* Negative screen for Hepatitis B surface (HBs) antigens, Hepatitis C Virus (HCV) antibodies, Hepatitis A Virus (HAV) antibodies and Human Immunodeficiency Virus (HIV) 1 and 2 antibodies
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participation in a clinical trial within 90 days prior to first drug administration
* Participants who have donated more than 500 milliliter (mL) of blood or who have lost significantly (more than 450 mL) blood within 90 days prior to first drug of administration
* Any surgical or medical condition, constitutes a risk or a contraindication for the participation of the participant in the study or that could interfere with the study objectives, conduct or evaluation
* History of surgery of the gastrointestinal tract
* Allergy
* Receipt of any prescription or non-prescription medication within 2 weeks before the first study drug administration
* Renal failure or renal dysfunction (creatinine clearance less than [<] 80 mL/minute) as assessed by using the estimated measure with the Cockcroft-Gault formula
* Known lack of participant compliance or inability to communicate or cooperate with the Investigator
* Considerable diet deviations from normal nutritional patterns
* Consumption of large quantities of methylxanthine-containing beverages (more than 600 milligram [mg] caffeine / day: one cup [240 mL] of coffee contains approx. 100 mg of caffeine, one cup of tea approximately 30 mg and one glass of cola approximately 20 mg caffeine)
* Consumption of grapefruit, orange, cranberry or juices of these fruits, 14 days prior to drug administration and during the study
* Legal incapacity or limited legal capacity
* Participants kept in detention
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4
Started | 10 | 10 | 10 | 10
Completed | 10 | 9 | 10 | 10
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4
Started | 10 | 9 | 10 | 10
Completed | 9 | 9 | 8 | 9
Not Completed | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1
Period: Treatment Period 4
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4
Started | 9 | 9 | 8 | 9
Completed | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.8 (9.8) | 23.9 (3.7) | 31.5 (8.3) | 25.7 (5.2) | 27.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 3 | 5 | 17
  Male | 4 | 7 | 7 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 10 | 10 | 40
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Metformin
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: The Pharmacokinetic (PK) analysis set included all participants who completed the trial with adequate trial medication compliance, without any relevant protocol violations with respect to factors likely to affect the comparability of PK results.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/ml)
Groups:
- Metformin-Gliclazide Combination: Participants received single oral dose of metformin 1000 mg and gliclazide 30 mg fixed combination tablet either in treatment period 1, 2, 3 or 4.
- Metformin and Gliclazide Separately: Participants received single oral dose of metformin 1000 mg and gliclazide 30 mg separately either in treatment period 1, 2, 3 or 4.
- Metformin: Participants received single oral dose of metformin 1000 mg either in treatment period 1, 2, 3 or 4.
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin
Number analyzed (Participants) | 35 | 35 | 35
nanogram*hour per milliliter (ng*h/ml) | 5033.8718 (1475.3418) | 6142.2821 (1848.4857) | 6090.7932 (1543.6463)
Statistical Analysis 1: Comparison: Metformin-Gliclazide Combination vs Metformin and Gliclazide Separately; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 81.4421, 90% CI 2-sided [75.2805 to 88.1079]
Statistical Analysis 2: Comparison: Metformin and Gliclazide Separately vs Metformin; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 102.2930, 90% CI 2-sided [97.8819 to 106.9028]
Statistical Analysis 3: Comparison: Metformin-Gliclazide Combination vs Metformin; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 81.0112, 90% CI 2-sided [74.8823 to 87.6417]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Gliclazide
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: The PK analysis set included all participants who completed the trial with adequate trial medication compliance, without any relevant protocol violations with respect to factors likely to affect the comparability of PK results.
Measure: Mean (Standard Deviation); unit: ng.h/ml
Groups:
- Gliclazide: Participants received single oral dose of gliclazide 30mg either in treatment period 1, 2, 3 or 4.
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Gliclazide
Number analyzed (Participants) | 35 | 35 | 35
ng.h/ml | 20707.7394 (8267.0653) | 20280.3103 (8219.1520) | 21205.2514 (7638.0877)
Statistical Analysis 1: Comparison: Metformin-Gliclazide Combination vs Metformin and Gliclazide Separately; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 102.2930, 90% CI 2-sided [97.8819 to 106.9028]
Statistical Analysis 2: Comparison: Metformin and Gliclazide Separately vs Gliclazide; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 105.7255, 90% CI 2-sided [101.1665 to 110.4900]
Statistical Analysis 3: Comparison: Metformin-Gliclazide Combination vs Gliclazide; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 96.7533, 90% CI 2-sided [92.5812 to 101.1135]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metformin
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin
Number analyzed (Participants) | 35 | 35 | 35
nanogram per milliliter (ng/ml) | 806.3895 (279.5063) | 1011.3941 (309.8136) | 977.2693 (262.4312)
Statistical Analysis 1: Comparison: Metformin-Gliclazide Combination vs Metformin and Gliclazide Separately; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 77.6923, 90% CI 2-sided [70.3830 to 85.7606]
Statistical Analysis 2: Comparison: Metformin and Gliclazide Separately vs Metformin; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 108.0819, 90% CI 2-sided [102.2370 to 114.2609]
Statistical Analysis 3: Comparison: Metformin-Gliclazide Combination vs Metformin; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 79.4367, 90% CI 2-sided [71.9633 to 87.6861]

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Gliclazide
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Gliclazide
Number analyzed (Participants) | 35 | 35 | 35
ng/ml | 972.168 (312.7305) | 892.6201 (259.7459) | 836.7239 (251.6451)
Statistical Analysis 1: Comparison: Metformin-Gliclazide Combination vs Metformin and Gliclazide Separately; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 108.0819, 90% CI 2-sided [102.2370 to 114.2609]
Statistical Analysis 2: Comparison: Metformin and Gliclazide Separately vs Gliclazide; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 93.6828, 90% CI 2-sided [88.6166 to 99.0386]
Statistical Analysis 3: Comparison: Metformin-Gliclazide Combination vs Gliclazide; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 115.3700, 90% CI 2-sided [109.1310 to 121.9658]

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Metformin
Description: AUC (0-inf) is defined as the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin
Number analyzed (Participants) | 35 | 35 | 35
ng*h/ml | 5313.3897 (1549.2688) | 6388.9849 (1857.6205) | 6341.5658 (1560.7170)
Statistical Analysis 1: Comparison: Metformin-Gliclazide Combination vs Metformin and Gliclazide Separately; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 82.6022, 90% CI 2-sided [76.5513 to 89.1314]
Statistical Analysis 2: Comparison: Metformin and Gliclazide Separately vs Metformin; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 101.8499, 90% CI 2-sided [97.8819 to 106.9028]
Statistical Analysis 3: Comparison: Metformin-Gliclazide Combination vs Metformin; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 81.0112, 90% CI 2-sided [74.8823 to 87.6417]

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Gliclazide
Description: as for outcome 5
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Gliclazide
Number analyzed (Participants) | 35 | 35 | 35
ng*h/ml | 21495.2343 (8358.3373) | 21120.6761 (8270.5092) | 22136.9988 (7687.4829)
Statistical Analysis 1: Comparison: Metformin-Gliclazide Combination vs Metformin and Gliclazide Separately; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 101.8499, 90% CI 2-sided [97.5947 to 106.2906]
Statistical Analysis 2: Comparison: Metformin and Gliclazide Separately vs Gliclazide; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 105.9150, 90% CI 2-sided [101.4900 to 110.5330]
Statistical Analysis 3: Comparison: Metformin-Gliclazide Combination vs Gliclazide; Test type: Equivalence — Bioequivalence boundaries of 80.000% to 125.00% were used; Geometric Least Squares Mean Ratio = 96.1619, 90% CI 2-sided [92.1443 to 100.3546]

7. Secondary Outcome: Apparent Volume of Distribution (Vz/f) of Metformin
Description: Vz/f was defined as apparent volume of distribution during terminal phase after non-intravenous administration.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin
Number analyzed (Participants) | 35 | 35 | 35
Milliliter | 1893618.4672 (1346880.1198) | 1414424.1926 (643556.2088) | 1489164.0229 (818767.0681)

8. Secondary Outcome: Apparent Volume of Distribution (Vz/f) of Gliclazide
Description: Vz/f was defined as apparent volume of distribution during terminal phase after non-intravenous administration.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Gliclazide
Number analyzed (Participants) | 35 | 35 | 35
Milliliter | 31636.8920 (7584.1651) | 32601.0115 (7057.8050) | 31413.9679 (6422.4920)

9. Secondary Outcome: Elimination Half Life (t1/2) of Metformin
Description: Elimination Half Life (t1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin
Number analyzed (Participants) | 35 | 35 | 35
Hours | 6.7151 (5.1372) | 5.9796 (2.8442) | 6.3048 (3.7114)

10. Secondary Outcome: Elimination Half Life (t1/2) of Gliclazide
Description: as for outcome 9
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Gliclazide
Number analyzed (Participants) | 35 | 35 | 35
Hours | 15.3086 (6.0231) | 15.4587 (5.6007) | 15.6222 (5.2904)

11. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Metformin
Description: CL/f was defined as apparent total clearance of the drug from plasma after oral administration.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter per Hour (mL/ h)
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin
Number analyzed (Participants) | 35 | 35 | 35
Milliliter per Hour (mL/ h) | 207132.8293 (70959.4296) | 170273.4024 (51108.0288) | 167260.5841 (39170.7306)

12. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Gliclazide
Description: CL/f was defined as apparent total clearance of the drug from plasma after oral administration.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Gliclazide
Number analyzed (Participants) | 35 | 35 | 35
mL/h | 1572.5246 (516.3724) | 1606.8952 (569.4811) | 1498.9932 (463.2158)

13. Secondary Outcome: Median Residence Time (MRT) for Metformin
Description: MRT is the average time that the molecules introduced into the body stays in the body.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin
Number analyzed (Participants) | 35 | 35 | 35
Hours | 8.3952 (3.0758) | 7.5836 (1.6807) | 7.7636 (2.0658)

14. Secondary Outcome: Median Residence Time (MRT) for Gliclazide
Description: MRT is the average time that the molecules introduced into the body stays in the body.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 28, 32, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Gliclazide
Number analyzed (Participants) | 35 | 35 | 35
Hours | 23.0593 (7.8010) | 24.4927 (7.7484) | 25.8590 (7.5834)

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 72
Population: The safety population included all participants who received at least 1 dose of the trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin | Gliclazide
Number analyzed (Participants) | 35 | 35 | 35 | 35
Participants
  TEAEs | 9 | 6 | 7 | 8
  SAEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 72
Description: The safety population included all participants who received at least 1 dose of the trial treatment.
Arm/Group | Metformin-Gliclazide Combination | Metformin and Gliclazide Separately | Metformin | Gliclazide
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 9/35 | 6/35 | 7/35 | 8/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin-Gliclazide Combination (N=35) | Metformin and Gliclazide Separately (N=35) | Metformin (N=35) | Gliclazide (N=35)
Elevated triglycerides (Investigations) | 1 | 3 | 2 | 0
High cholesterol (Investigations) | 0 | 0 | 1 | 0
Elevated alanine aminostrasferase (Investigations) | 1 | 0 | 4 | 1
Elevated aspartate aminotrasferase (Investigations) | 1 | 0 | 5 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 2 | 5 | 7
Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Infectious gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Wound in the left submaxillary region (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urinary infection (Infections and infestations) | 1 | 0 | 0 | 0
Urethritis (Infections and infestations) | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT03467945/SAP_000.pdf
  • Study Protocol (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03467945/Prot_001.pdf